CLINICAL TRIAL: NCT07160361
Title: Exploration of Postoperative Adjuvant Therapy for Hepatocellular Carcinoma Patients With Positive Tumor Budding
Brief Title: Exploration of Postoperative Adjuvant Therapy for HCC Patients With Positive TB
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Collaborators: First Affiliated Hospital Xi'an Jiaotong University (Other); Shaanxi Provincial People's Hospital (Other); Affiliated Hospital of Qinghai University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XJTUSAH-TB-Z008
Record Dates: First submitted 2025-08-30; First posted 2025-09-08 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-08

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib; Losartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lenvatinib + losartan treatment group (Experimental)
  Interventions: Drug: Lenvatinib + losartan

INTERVENTIONS:
Drug: Lenvatinib + losartan — Patients will receive a combination of lenvatinib and losartan at the same time after surgery for treatment cycles once daily (lenvatinib and losartan).
  Adjuvant therapy will be started within 2-6 weeks after surgery for a period of time to evaluate the effect of different treatment regimens on reducing tumor recurrence and improving survival.
  lenvatinib: orally once daily according to standard dosing guidelines, starting postoperatively.
  losartan: 50mg losartan potassium tablets orally once daily starting postoperatively.

SUMMARY:
Hepatocellular carcinoma (HCC) is one of the most common types of primary liver cancer worldwide, characterized by complex and variable disease progression and significant treatment challenges. Among HCC patients, tumor budding (TB) is associated with a high risk of postoperative recurrence, significantly impacting patient prognosis. Even in the current HCC pathological diagnosis "gold standard" of MVI-negative patients, TB retains excellent prognostic predictive value. TB cells reside within the peritumoral stroma, where dense collagen fibers restrict the efficacy of therapeutic agents including chemotherapy, immunotherapy, and targeted therapies, making it difficult for single-agent treatments to effectively eliminate TB. Therefore, specific treatment strategies should be considered for TB-positive patients to improve survival outcomes and reduce the risk of tumor recurrence. To address this clinical challenge, this study aims to clarify the prognostic impact of combining collagen degradation therapy with targeted therapy in TB-positive HCC patients. Through a single-arm trial (postoperative targeted therapy + collagen degradation therapy), investigators explore the clinical efficacy and prognostic indicators of this combination approach, seeking the optimal treatment strategy for TB-positive HCC patients. Collagen degradation therapy facilitates drug delivery to tumor-bottle lesions by degrading collagen barriers, while targeted therapy specifically intervenes against cancer cells. Their combination holds promise for synergistic effects and enhanced therapeutic outcomes. This study aims to preliminarily assess the impact of this dual approach on prognosis, providing evidence for personalized treatment strategies. The findings of this research hold promise for delivering new breakthroughs in the treatment of TB-positive HCC patients, improving their quality of life and survival rates, and providing robust support for future clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age is ≥18 years old, male or female;
* Histologically confirmed as hepatocellular carcinoma without metastasis;
* Tumor budding is positive
* Life expectancy of at least 12 weeks;

Exclusion Criteria:

* Hepatocellular carcinoma that cannot be surgically resected
* Received radiotherapy, chemotherapy, targeted therapy, immunotherapy, etc. before surgery
* Pregnant or lactating women
* Subjects with other malignant tumors;
* Subjects who are considered unsuitable to participate in this cohort study by the investigator;
* Subjects who refuse to enroll or do not sign the informed consent form;
* Subjects with incomplete medical record information (including gender, age, diagnostic information, imaging (and) or pathological diagnosis results, other demographic data, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Relapse rate within 2 years | 2 years